CLINICAL TRIAL: NCT06382519
Title: Thalidomide Therapy for Very Early Onset Inflammatory Bowel Disease
Brief Title: Thalidomide Therapy for VEOIBD
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Ying HUANG, Head of gastroenterology department, Children's Hospital of Fudan University
Other Study IDs: Thal in VEOIBD
Record Dates: First submitted 2024-04-11; First posted 2024-04-24 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Thalidomide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sample, stool samples and biopsy samples during endoscopy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Thalidomide — thalidomide, dose 1.5-2.5mg/kg.d, orally taken before bedtime.

SUMMARY:
This is a single center, observational study to investigate the clinical outcomes of thalidomide treatment for very early onset inflammatory bowel disease

DETAILED DESCRIPTION:
Very early onset inflammatory bowel disease (VEOIBD) refers to IBD diagnosed before 6 years of age. VEOIBD comprises a distinct subset of pediatric IBD characterized by stronger genetic predisposition, predominant colonic involvement, more extensive inflammation, more severe course, and peculiar response to treatments. Previous studies have been demonstrated that thalidomide, an oral molecule with immunomodulatory, antiangiogenic, and TNF-suppressing properties, is an effective and safe treatment for adults and children with IBD refractory to conventional therapies. This study is aimed to evaluate the efficacy and tolerance of thalidomide in VEOIBD.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with inflammatory bowel disease
* disease onset less than 6 years old
* Pediatric Crohn's disease Activity Index (PCDAI)>30 or Pediatric Ulcerative Colitis Activity Index (PUCAI)>35
* patients and their legal guardians were willing to receive thalidomide treatment and participate in this study.

Exclusion Criteria:

* liver dysfunction
* allergy to thalidomide
* with Neuropathy
* with thrombosis
* thalidomide treatment in the previous 30 days
* biologics treatment in the previous 8 weeks
* not suitable participated in this study

Ages: 28 Days to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children diagnosed with very early onset inflammatory bowel disease who were seen at the Children's hospital of Fudan university who met the inclusion and exclusion criteria would be enrolled in this study.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
endoscopic response rate | week 52
  The Simple Endoscopic Score for Crohn Disease decreased 50% compared with baseline OR Mayo score 0-1 (higher scores mean a worse outcome)

SECONDARY OUTCOMES:
clinical response rate | week8, week26, week52
  Inflammatory bowel disease mainly contains Crohn's disease and ulcerative colitis. If the patient was diagnosed with Crohn's disease, we use the Pediatric Crohn's disease Activity Index score to evaluate the clinical response, which is defined as Pediatric Crohn's disease Activity Index decreased more than 12.5 compared with baseline. If the patient was diagnosed with ulcerative colitis, we use the Pediatric Ulcerative Colitis Activity Index score to evaluate the clinical response, which is defined as Pediatric Ulcerative Colitis Activity Index score decreased more than 20 compared with baseline. The Pediatric Crohn's disease Activity Index score varies from 0 to 100 and the Pediatric Ulcerative Colitis Activity Index score varies from 0 to 85 (higher scores mean a worse outcome).
biomarker remission rate | week8, week26, week52
  biomarker remission is defined as not only C-reactive protein less than 8mg/L, but also fecal calprotectin less than 100ug/g.
growth development | week52
  weight and height Z score (higher scores mean a better outcome)
clinical remission rate with steroid-free | week26
  If the patient was diagnosed with Crohn's disease, this outcome is defined as the Pediatric Crohn's disease Activity Index score less than 10 without steroid treatment. If the patient was diagnosed with ulcerative colitis, this outcome is defined as the Pediatric Ulcerative Colitis Activity Index score less than 10 without steroid treatment.
adverse event | within one year
  The rate of the potential adverse events were monitored during the intervention.
treatment persistence | within one year
  the time between the start and the last dose of thalidomide

CONTACTS AND LOCATIONS:
Overall Officials: Ying Huang, Principal Investigator — Children's Hospital of Fudan University
Locations (1):
- Lin Wang, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided